CLINICAL TRIAL: NCT04345289
Title: Efficacy and Safety of Treatment With Convalescent Plasma for Adults With COVID-19 Pneumonia. A Double-blinded, Randomized, Multicenter Placebo-controlled Trial
Brief Title: Efficacy and Safety of Novel Treatment Options for Adults With COVID-19 Pneumonia
Acronym: CCAP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB advise due to high probability of futility
Sponsor: Thomas Benfield (Other)
Responsible Party: Sponsor-Investigator, Thomas Benfield, Professor, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25032020; 2020-001367-88 (EudraCT Number)
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: COVID; Corona Virus Infection; Viral Pneumonia
MeSH Terms: conditions — Coronavirus Infections; Pneumonia, Viral

STUDY DESIGN:
Intervention Model Description: Adaptive multi-arm trial comparing convalescent plasma against control group. Interim analyses are included at 300 and 700 included participants to compare the effect and safety of the experimental treatment to control (placebo). The results of the interim analyses are used to decide if the treatments should be discontinued due to either futility or harm. The study is discontinued if either of the predefined stopping criteria are met.
  Additional experimental treatments may be added as they become available. Any efficacious treatment identified in this or any other high-quality RCT may become the new SOC after consensus by national and international societies, and, thus, the control arm will change accordingly and in parallel.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both convalescent plasma and placebo will be administered via a colored intravenous line with a colored sleeve disguising the fluid bag.
  In order to achieve blinding of participants and treating personnel, patients randomized to active treatment will also receive placebo treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Convalescent plasma (Active Comparator): Will receive active treatment with convalescent anti-SARS-CoV-2 plasma (600 ml) as a single dose iv infusion in addition to standard care.
  Interventions: Biological: Convalescent anti-SARS-CoV-2 plasma
- Infusion placebo (Placebo Comparator): Will receive placebo treatment with saline 0.9% (2 x 300 ml) as an iv single dose infusion in addition to standard care.
  Interventions: Other: Infusion placebo

INTERVENTIONS:
Biological: Convalescent anti-SARS-CoV-2 plasma — Single infusion of convalescent anti-SARS-CoV-2 plasma (2 x 300 mL)
  Other Names: Convalescent plasma
  Arms: Convalescent plasma
Other: Infusion placebo — Saline 0.9% (600 ml) as an iv single dose infusion
  Arms: Infusion placebo

SUMMARY:
CCAP is an investigator-initiated multicentre, randomized, double blinded, placebo-controlled trial, which aims to assess the safety and efficacy of treatment with convalescent plasma for patients with moderate-severe COVID-19.

Participants will be randomized 2:1 to two parallel treatment arms: Convalescent plasma, and intravenous placebo.

Primary outcome is a composite endpoint of all-cause mortality or need of invasive mechanical ventilation up to 28 days.

DETAILED DESCRIPTION:
The study is a randomized, double blinded, placebo-controlled, multicenter study with two parallel treatment arms consisting of either convalescent plasma or intravenous placebo. We plan to enroll a total of 1100 patients yielding a statistical power of 80 % to show a 30% relative reduction in risk of mechanical ventilation or death at day 28. Patients with confirmed COVID-19 infection and signs compatible with pneumonia will be enrolled in the study. The participants will be randomized 2:1 to the parallel treatment arms, and receive either single dose infusion treatment.

The primary outcome is a composite endpoint of all-cause mortality or need of invasive mechanical ventilation up to 28 days. Interim analysis will be performed frequently.

As new knowledge of treatment options for COVID-19 have emerged, the treatment arms including sarilumab, baricitininb, hydroxychloroquine and oral placebo have been terminated.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Confirmed COVID-19 infection by presence of SARS-CoV-2 nucleic acid by polymerase chain reaction (PCR)
* Evidence of pneumonia given by at least one of the following: SpO2 ≤93% on ambient air or PaO2/FiO2 <300 mmHg/40 kPa OR Radiographic findings compatible with COVID-19 pneumonia
* For women of childbearing potential: Negative pregnancy test and willingness to use contraceptive (consistent with local regulations) during study period
* Signed Informed Consent Form by any patient capable of giving consent, or, when the patient is not capable of giving consent, by his or her legal/authorized representatives

Exclusion Criteria:

* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatment
* Participating in other drug clinical trials (participation in COVID-19 antiviral trials may be permitted if approved by sponsor)*
* Pregnant or breastfeeding, positive pregnancy test in a pre-dose examination
* Any serious medical condition or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
All-cause mortality or need of invasive mechanical ventilation | 28 days
  Composite outcome

SECONDARY OUTCOMES:
Frequency of adverse events | 90 days
  Number of participants with adverse events with possible relation to study drug
Frequency of severe adverse events | 90 days
  Number of participants with serious adverse events according to International Council of Harmonisation-Good Clinical Practice (ICH-GCP) guidelines
Time to improvement of at least 2 categories relative to baseline on a 7-category ordinal scale of clinical status | 90 days
  Number of days to improvement of at least 2 categories relative to baseline on the ordinal scale. Categories are as follows: Death; Hospitalized, in intensive care requiring Extracorporeal Membrane Oxygenation (ECMO) or mechanical ventilation; Hospitalized, on non-invasive ventilation or high-flow oxygen device; Hospitalized, requiring supplemental oxygen; Hospitalized, not requiring supplemental oxygen; Not hospitalized, limitation on activities and/or requiring home oxygen; Not hospitalized, no limitations on activities
Ventilator-free days | 28 days
  Number of days without mechanical ventilation
Organ failure-free days | 28 days
  Number of days without organ-failure
Duration of ICU stay | 90 days
  Number of days in ICU
Mortality rate | 7, 14, 21, 28 and 90 days
  Number of deaths by any cause
Length of hospital stay | 90 days
  Days from the date of hospital admission for COVID-19 to the date of discharge
Duration of supplemental oxygen | 90 days
  Days requiring supplement oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Hansen, MD, Study Director — Hvidovre University Hospital; Simone Bastrup Israelsen, MD, Study Director — Hvidovre University Hospital; Louise Thorlacius-Ussing, MD, Study Director — Hvidovre University Hospital; Karen Brorup Heje Pedersen, MD, Study Director — Hvidovre University Hospital; Clara Clausen, MD, Study Director — Hvidovre University Hospital; Michaela Tinggaard, MD, Study Director — Hvidovre University Hospital; Nichlas Hovmand, MD, Study Director — Hvidovre University Hospital
Locations (12):
- Denmark (12):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Herlev Gentofte Hospital, Herlev
  - Herning Hospital, Herning
  - Nordsjællands Hospital, Hillerød
  - Hvidovre Hospital, Hvidovre
  - Kolding Hospital, Kolding
  - Odense University Hospital, Odense
  - Roskilde Hospital, Roskilde
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Infection prevention and control in the context of coronavirus disease 2019 (COVID-19): a living guideline [Internet]. Geneva: World Health Organization; 2022 Apr 25-. Available from http://www.ncbi.nlm.nih.gov/books/NBK581594/ PMID 35767666
- [Background] Cameron MJ, Bermejo-Martin JF, Danesh A, Muller MP, Kelvin DJ. Human immunopathogenesis of severe acute respiratory syndrome (SARS). Virus Res. 2008 Apr;133(1):13-9. doi: 10.1016/j.virusres.2007.02.014. Epub 2007 Mar 19. PMID 17374415
- [Background] Matthay MA, Ware LB, Zimmerman GA. The acute respiratory distress syndrome. J Clin Invest. 2012 Aug;122(8):2731-40. doi: 10.1172/JCI60331. Epub 2012 Aug 1. PMID 22850883
- [Background] Channappanavar R, Perlman S. Pathogenic human coronavirus infections: causes and consequences of cytokine storm and immunopathology. Semin Immunopathol. 2017 Jul;39(5):529-539. doi: 10.1007/s00281-017-0629-x. Epub 2017 May 2. PMID 28466096
- [Background] Li Y, Chen M, Cao H, Zhu Y, Zheng J, Zhou H. Extraordinary GU-rich single-strand RNA identified from SARS coronavirus contributes an excessive innate immune response. Microbes Infect. 2013 Feb;15(2):88-95. doi: 10.1016/j.micinf.2012.10.008. Epub 2012 Oct 30. PMID 23123977
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Devaux CA, Rolain JM, Colson P, Raoult D. New insights on the antiviral effects of chloroquine against coronavirus: what to expect for COVID-19? Int J Antimicrob Agents. 2020 May;55(5):105938. doi: 10.1016/j.ijantimicag.2020.105938. Epub 2020 Mar 12. PMID 32171740
- [Background] Luke TC, Kilbane EM, Jackson JL, Hoffman SL. Meta-analysis: convalescent blood products for Spanish influenza pneumonia: a future H5N1 treatment? Ann Intern Med. 2006 Oct 17;145(8):599-609. doi: 10.7326/0003-4819-145-8-200610170-00139. Epub 2006 Aug 29. PMID 16940336
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Taylor PC, Keystone EC, van der Heijde D, Weinblatt ME, Del Carmen Morales L, Reyes Gonzaga J, Yakushin S, Ishii T, Emoto K, Beattie S, Arora V, Gaich C, Rooney T, Schlichting D, Macias WL, de Bono S, Tanaka Y. Baricitinib versus Placebo or Adalimumab in Rheumatoid Arthritis. N Engl J Med. 2017 Feb 16;376(7):652-662. doi: 10.1056/NEJMoa1608345. PMID 28199814
- [Background] Wu D, Yang XO. TH17 responses in cytokine storm of COVID-19: An emerging target of JAK2 inhibitor Fedratinib. J Microbiol Immunol Infect. 2020 Jun;53(3):368-370. doi: 10.1016/j.jmii.2020.03.005. Epub 2020 Mar 11. PMID 32205092
- [Background] Stebbing J, Phelan A, Griffin I, Tucker C, Oechsle O, Smith D, Richardson P. COVID-19: combining antiviral and anti-inflammatory treatments. Lancet Infect Dis. 2020 Apr;20(4):400-402. doi: 10.1016/S1473-3099(20)30132-8. Epub 2020 Feb 27. No abstract available. PMID 32113509
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Cunningham AC, Goh HP, Koh D. Treatment of COVID-19: old tricks for new challenges. Crit Care. 2020 Mar 16;24(1):91. doi: 10.1186/s13054-020-2818-6. No abstract available. PMID 32178711
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Soo YO, Cheng Y, Wong R, Hui DS, Lee CK, Tsang KK, Ng MH, Chan P, Cheng G, Sung JJ. Retrospective comparison of convalescent plasma with continuing high-dose methylprednisolone treatment in SARS patients. Clin Microbiol Infect. 2004 Jul;10(7):676-8. doi: 10.1111/j.1469-0691.2004.00956.x. PMID 15214887
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Zou L, Ruan F, Huang M, Liang L, Huang H, Hong Z, Yu J, Kang M, Song Y, Xia J, Guo Q, Song T, He J, Yen HL, Peiris M, Wu J. SARS-CoV-2 Viral Load in Upper Respiratory Specimens of Infected Patients. N Engl J Med. 2020 Mar 19;382(12):1177-1179. doi: 10.1056/NEJMc2001737. Epub 2020 Feb 19. No abstract available. PMID 32074444
- [Background] Zhang Y, Li J, Zhan Y, Wu L, Yu X, Zhang W, Ye L, Xu S, Sun R, Wang Y, Lou J. Analysis of serum cytokines in patients with severe acute respiratory syndrome. Infect Immun. 2004 Aug;72(8):4410-5. doi: 10.1128/IAI.72.8.4410-4415.2004. PMID 15271897
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Pelechas E, Voulgari PV, Drosos AA. Clinical evaluation of the safety, efficacy and tolerability of sarilumab in the treatment of moderate to severe rheumatoid arthritis. Ther Clin Risk Manag. 2019 Sep 4;15:1073-1079. doi: 10.2147/TCRM.S167452. eCollection 2019. PMID 31564885
- [Background] Vincent MJ, Bergeron E, Benjannet S, Erickson BR, Rollin PE, Ksiazek TG, Seidah NG, Nichol ST. Chloroquine is a potent inhibitor of SARS coronavirus infection and spread. Virol J. 2005 Aug 22;2:69. doi: 10.1186/1743-422X-2-69. PMID 16115318
- [Background] Klumperman J, Locker JK, Meijer A, Horzinek MC, Geuze HJ, Rottier PJ. Coronavirus M proteins accumulate in the Golgi complex beyond the site of virion budding. J Virol. 1994 Oct;68(10):6523-34. doi: 10.1128/JVI.68.10.6523-6534.1994. PMID 8083990
- [Background] Gay B, Bernard E, Solignat M, Chazal N, Devaux C, Briant L. pH-dependent entry of chikungunya virus into Aedes albopictus cells. Infect Genet Evol. 2012 Aug;12(6):1275-81. doi: 10.1016/j.meegid.2012.02.003. Epub 2012 Feb 20. PMID 22386853
- [Background] multicenter collaboration group of Department of Science and Technology of Guangdong Province and Health Commission of Guangdong Province for chloroquine in the treatment of novel coronavirus pneumonia. [Expert consensus on chloroquine phosphate for the treatment of novel coronavirus pneumonia]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Mar 12;43(3):185-188. doi: 10.3760/cma.j.issn.1001-0939.2020.03.009. Chinese. PMID 32164085
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Jaki T, Wason JMS. Multi-arm multi-stage trials can improve the efficiency of finding effective treatments for stroke: a case study. BMC Cardiovasc Disord. 2018 Nov 27;18(1):215. doi: 10.1186/s12872-018-0956-4. PMID 30482176
- [Background] Cordon-Cardo C, Lloyd KO, Finstad CL, McGroarty ME, Reuter VE, Bander NH, Old LJ, Melamed MR. Immunoanatomic distribution of blood group antigens in the human urinary tract. Influence of secretor status. Lab Invest. 1986 Oct;55(4):444-54. PMID 2429066
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Distler P. ISBT 128: a global information standard. Cell Tissue Bank. 2010 Nov;11(4):365-73. doi: 10.1007/s10561-010-9196-2. Epub 2010 Jul 21. PMID 20652420
- [Background] Clegg DO, Dietz F, Duffy J, Willkens RF, Hurd E, Germain BF, Wall B, Wallace DJ, Bell CL, Sleckman J. Safety and efficacy of hydroxychloroquine as maintenance therapy for rheumatoid arthritis after combination therapy with methotrexate and hydroxychloroquine. J Rheumatol. 1997 Oct;24(10):1896-902. PMID 9330929
- [Background] Middelburg RA, Van Stein D, Zupanska B, Uhrynowska M, Gajic O, Muniz-Diaz E, Galvez NN, Silliman CC, Krusius T, Wallis JP, Vandenbroucke JP, Briet E, Van Der Bom JG. Female donors and transfusion-related acute lung injury: A case-referent study from the International TRALI Unisex Research Group. Transfusion. 2010 Nov;50(11):2447-54. doi: 10.1111/j.1537-2995.2010.02715.x. PMID 20529001
- [Background] Lamb YN, Deeks ED. Sarilumab: A Review in Moderate to Severe Rheumatoid Arthritis. Drugs. 2018 Jun;78(9):929-940. doi: 10.1007/s40265-018-0929-z. PMID 29931592
- [Background] Pocock SJ, Ariti CA, Collier TJ, Wang D. The win ratio: a new approach to the analysis of composite endpoints in clinical trials based on clinical priorities. Eur Heart J. 2012 Jan;33(2):176-82. doi: 10.1093/eurheartj/ehr352. Epub 2011 Sep 6. PMID 21900289
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Rodriguez-Morales AJ, Cardona-Ospina JA, Gutierrez-Ocampo E, Villamizar-Pena R, Holguin-Rivera Y, Escalera-Antezana JP, Alvarado-Arnez LE, Bonilla-Aldana DK, Franco-Paredes C, Henao-Martinez AF, Paniz-Mondolfi A, Lagos-Grisales GJ, Ramirez-Vallejo E, Suarez JA, Zambrano LI, Villamil-Gomez WE, Balbin-Ramon GJ, Rabaan AA, Harapan H, Dhama K, Nishiura H, Kataoka H, Ahmad T, Sah R; Latin American Network of Coronavirus Disease 2019-COVID-19 Research (LANCOVID-19). Electronic address: https://www.lancovid.org. Clinical, laboratory and imaging features of COVID-19: A systematic review and meta-analysis. Travel Med Infect Dis. 2020 Mar-Apr;34:101623. doi: 10.1016/j.tmaid.2020.101623. Epub 2020 Mar 13. PMID 32179124
- [Derived] Thorlacius-Ussing L, Brooks PT, Nielsen H, Jensen BA, Wiese L, Saekmose SG, Johnsen S, Gybel-Brask M, Johansen IS, Bruun MT, Staerke NB, Ostergaard L, Erikstrup C, Ostrowski SR, Homburg KM, Georgsen J, Mikkelsen S, Sandholdt H, Leding C, Hovmand N, Clausen CL, Tinggaard M, Pedersen KBH, Iversen KK, Tingsgard S, Israelsen SB, Benfield T. A randomized placebo-controlled trial of convalescent plasma for adults hospitalized with COVID-19 pneumonia. Sci Rep. 2022 Sep 30;12(1):16385. doi: 10.1038/s41598-022-19629-z. PMID 36180450